CLINICAL TRIAL: NCT01489514
Title: Evaluation of Allergenicity of Hypoallergenic Peanut Product in Peanut Allergic Subjects.
Acronym: peanut
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Investigator, University of North Carolina, Chapel Hill
Other Study IDs: IRB# 10-0851
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Peanut Allergy
Keywords: peanut allergy; hypoallergenic peanut extracts; epicutaneous skin prick testing
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venipuncture for 30mL of blood taken for measurement of peanut IgE.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peanut allergic subjects
  Interventions: Other: Epicutaneous skin prick testing

INTERVENTIONS:
Other: Epicutaneous skin prick testing — Epicutaneous skin prick testing will be performed utilizing the following extracts:
  1. Histamine control purchased from Greer.
  2. Saline control purchased from Greer.
  3. Standard Peanut Extract purchased from Greer.
  4. Sterile extract prepared from Trypsin and Chymotrypsin treated peanuts. This is prepared by North Carolina A & T.
  5. Sterile extract prepared from roasted & blanched but untreated peanuts. This is prepared by North Carolina A & T.
  6. Sterile extract prepared from peanuts (no blanching, no enzyme). This is prepared by North Carolina A & T. This is not classified as a drug and is
  7. Sterile extract containing peanuts treated with 0.2% inactivated a-chymotrypsin and trypsin as an enzyme negative control.
  8. Sterile extracts containing peanuts that have been treated with alcalase

SUMMARY:
This is a proof of concept study to determine the safety and allergenicity of hypoallergenic peanut product extract as compared to standard peanut extract in an adult population with known peanut allergy. This will be assessed by epicutaneous skin prick testing. The hypothesis is that subjects with previously diagnosed peanut allergy will have less epicutaneous reactions to the hypoallergenic peanut product extract.

DETAILED DESCRIPTION:
Peanut allergic volunteers will be identified by positive skin prick test to peanut (peanut extract obtained from Greer laboratories). The peanut extract to be used is FDA approved and is routinely used in confirming a diagnosis of peanut allergy. Serum Total IgE and peanut-specific IgE will be measured for assessment of atopy in general and confirmation of Peanut allergy respectively. Only patients with positive skin test to peanut will enrolled into the study.

Allergic volunteers will be asked to abstain from taking any antihistamines (H1 or H2) during the 3 days prior to the skin testing.

Testing day

1. Obtain informed consent
2. Obtain medical history, list of current medications
3. Vital signs.
4. Obtain urine pregnancy test if applicable
5. Perform partial physical exam (PE) to include, ENT, Eyes, Neck, Respiratory, Cardiac and Skin with focus mainly on lungs to rule out bronchospasm/asthma exacerbation.
6. Epicutaneous skin prick testing with histamine and saline control, standard peanut extract will be done on all subjects (Total skin prick=3). Those subjects who qualify for the study (test positive to standard peanut extract) will then undergo skin prick testing with standard histamine control, standard saline control, hypoallergenic (Trypsin+Chymotrypsin treated) extract, extract from blanched untreated (no enzyme) peanuts, non-blanched untreated extracts, and peanuts treated with 0.2% inactivated a-chymotrypsin and trypsin as an enzyme control. A second set of skin testing reagents may used these reagents have been treated with alcalase. Skin testing will be read at 15 minutes. A positive test is defined as ≥ 3mm wheal compared to saline control. DermaPIK device will be used for this skin prick testing.
7. Obtain blood samples One time 20ml collection for determination of total IgE, peanut specific IgE in peanut allergic individuals only.

Physical Exams will be performed by a study physician. Procedures such as skin testing, vital signs, venipuncture, will be done by a study coordinator, qualified nurse or technical staff. Clinical labs (Serum IgE and Peanut-specific IgE) will be processed at Labcorp Inc in Burlington, NC.

Recording of Skin Test results: Skin test reactions will be traced onto clear cellophane tape from which measurements will be obtained. This tape will be affixed to a subject's visit record but not their personal medical record.

Excess samples remaining after completion of analyses for this study will be stored in the CEMALB Repository (IRB #05-2528) and all participants will be asked to sign the Repository consent form. Failure to consent to the repository will not result in exclusion from the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Specific allergy to peanut confirmed by positive immediate skin test response.
2. Oxygen saturation of > 94 % at baseline
3. Blood pressure within the following parameters (Systolic between 140 - 90, Diastolic between 90-60 mm Hg)
4. Must be willing and medically able to withhold antihistamine treatment (both H1 and H2) for 3 days prior to starting study medication, and for the duration of the treatment period. Any subject will be told to resume their antihistamine treatment if symptoms require resuming medication.

Exclusion Criteria:

1. Any chronic medical condition including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, chronic thyroid disease, kidney disease or coagulation defects. Asthma is not an exclusion criterion.
2. Asthmatic patients must be on a stable regimen of asthma therapy which has not changed in the past month prior to entrance into the study.
3. Asthmatic or allergic non-asthmatic patients must not be on leukotriene receptor antagonists, as this may potentially interfere with epicutaneous skin testing and in vitro allergen-induced leukotriene production
4. Pregnancy or nursing a baby. As this is a phase I study, the potential risk to a fetus cannot be justified.
5. Children will not be included in this study as the potential risk to a growing child cannot be justified.
6. Adults age 66 and older are excluded as the potential for concomitant illness in this population increases the risk for confounding the data.
7. Known vagal response to venipuncture
8. Hypertension, classified as a systolic blood pressure of equal to or greater than 140, and a diastolic blood pressure equal to or greater than 90.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty (30) adult subjects with history of peanut allergy, with or without asthma will be recruited. All participants will be adults ages 18-65. There will no gender or ethnic restrictions.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Size of wheal with epicutaneous testing using non-hypoallergenic extracts. | 20 minutes
  Size of wheal for hypoallergenic extracts will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Yu, J; Hernandez, M; Li, H; Goktepe, I; Robinette, C; Auerbach, A; Peden, D; Ahmedna, M. Allergenicity of roasted peanuts treated with a non-human digestive protease. Food Research International 2015 March; 69: 341-47. doi:10.1016/j.foodres.2015.01.007